CLINICAL TRIAL: NCT02156765
Title: China Atrial Fibrillation Screening in Acute Ischemic Stroke Patients
Acronym: CRIST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: yongjun wang (Other Government)
Responsible Party: Sponsor-Investigator, yongjun wang, vice president of Tiantan Hospital, Ministry of Science and Technology of the People´s Republic of China
Organization: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Other Study IDs: TTYY-20140410
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Atrial Fibrillation; Screening; Stroke patients
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Three purpose of this study:

1. Increase diagnosis rate and formulate the flow of diagnosis and treatment of AF in ischemic stroke patients;
2. Evaluation on specificity and sensitivity of STAF score;
3. Analyze the pathogenesis of ischemic stroke and risk factors and establish clinical database and sample database of ischemic stroke.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Hospitalized patients with ischemic stroke that are diagnosed definitely;
2. Age ≥ 18 years;
3. Within 7 days after the onset of diseases;
4. Signed the consent informed form.

Exclusion criteria:

1. Patients with noncerebrovascular diseases that are diagnosed definitely;
2. Silent cerebral infarction (CI) without symptoms and signs;
3. Those refuse to sign the consent informed form of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients with ischemic stroke that are diagnosed definitely;
2. Age ≥ 18 years;
3. Within 7 days after the onset of diseases;
4. Signed the consent informed form.

Exclusion Criteria:

1. Patients with noncerebrovascular diseases that are diagnosed definitely;
2. Silent cerebral infarction (CI) without symptoms and signs;
3. Those refuse to sign the consent informed form of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with ischemic stroke that are diagnosed definitely
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Accumulated detection rate of AF | 1.5 year
  ECG was monitored for all patients enrolled in a single center for consecutive 6 days

CONTACTS AND LOCATIONS:
Overall Officials: yongjun wang, doctor, Principal Investigator — Tiantan Hospital
Locations (1):
- Beijing Stroke Association, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Ay H, Furie KL, Singhal A, Smith WS, Sorensen AG, Koroshetz WJ. An evidence-based causative classification system for acute ischemic stroke. Ann Neurol. 2005 Nov;58(5):688-97. doi: 10.1002/ana.20617. PMID 16240340
- [Derived] Li SY, Yang XM, Zhao XQ, Liu LP, Wang YL, Jiang Y, Wang YJ. Newly detected atrial fibrillation is associated with cortex-involved ischemic stroke. Chin Med J (Engl). 2019 Sep 5;132(17):2053-2058. doi: 10.1097/CM9.0000000000000390. PMID 31403970
- [Derived] Yang X, Li S, Zhao X, Liu L, Jiang Y, Li Z, Wang Y, Wang Y. Atrial fibrillation is not uncommon among patients with ischemic stroke and transient ischemic stroke in China. BMC Neurol. 2017 Dec 4;17(1):207. doi: 10.1186/s12883-017-0987-y. PMID 29202727